CLINICAL TRIAL: NCT03243864
Title: : Pharmacokinetics of Ceftazidime-Avibactam in Critically Ill Patients With Renal Failure Requiring Continuous Venovenous Hemodiafiltration
Brief Title: Study of Ceftazidime-Avibactam Blood Concentrations in Intensive Care Unit Patients With Renal Failure Requiring Continuous Dialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 866
Record Dates: First submitted 2017-08-01; First posted 2017-08-09 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Renal Failure; Bacterial Infections; Critical Illness
MeSH Terms: conditions — Renal Insufficiency; Bacterial Infections; Critical Illness | interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood, plasma, effluent fluid from dialysis machine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ceftazidime and Avibactam: Ceftazidime-avibactam pharmacokinetic monitoring
  Interventions: Drug: Ceftazidime-avibactam

INTERVENTIONS:
Drug: Ceftazidime-avibactam — Patients will be started on 2.5 gm IV every 8 hours
  Other Names: Avycaz

SUMMARY:
The study's primary objective is to determine plasma and dialysis fluid concentrations in patients prescribed ceftazidime-avibactam as the standard treatment for their infection and requiring continuous venovenous hemodiafiltration (CVVHDF) as part of the standard treatment for acute or chronic renal failure. Secondarily, the study will evaluate the pharmacokinetics of ceftazidime-avibactam in these patients on CVVHDF. The study will also determine if the prescribed dose meets pharmacodynamic targets.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Patients requiring continuous renal replacement therapy (CRRT) due to acute or chronic renal failure
* documented or suspected infection requiring a prescription for ceftazidime-avibactam

Exclusion Criteria:

* Patients on CRRT < 24 hours
* Patients on ceftazidime-avibactam < 24 hours
* Patients unable to remain on CRRT for 32 hours continuously without clotting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2020-03-21 (Estimated); Study Completion 2020-10-21 (Estimated)

PRIMARY OUTCOMES:
Ceftazidime plasma concentrations | At hours post dose: 0, 2, 3, 4, 6, 8 on or after Day 2 of therapy (i.e. during the fourth dose)
  mg/L
Avibactam plasma concentrations | At hours post dose: 0, 2, 3, 4, 6, 8 on or after Day 2 of therapy (i.e. during the fourth dose)
  mg/L
Ceftazidime effluent concentrations | At hours post dose: 0, 2, 3, 4, 6, 8 on or after Day 2 of therapy (i.e. during the fourth dose)
  mg/L
Avibactam effluent concentrations | At hours post dose: 0, 2, 3, 4, 6, 8 on or after Day 2 of therapy (i.e. during the fourth dose)
  mg/L

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | At hours post dose: 0, 2, 3, 4, 6, 8 on or after Day 2 of therapy (i.e. during the fourth dose)
  mg/L
Number of participants with adverse effects as a measure of safety | Days 1-30
  Measure of safety
Minimum plasma concentration (Cmin) | At hours post dose: 0, 2, 3, 4, 6, 8 on or after Day 2 of therapy (i.e. during the fourth dose)
  mg/L
Half-life (t1/2) | 8-hours
  hours
Clearance (Cl) | 8-hours
  L/hr
AUC 0 to 8 hours | 8-hours
  mg*hr/L
Sieving Coefficient | 8-hours
  SC

CONTACTS AND LOCATIONS:
Overall Officials: Christina Rose, Pharm.D., Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No